CLINICAL TRIAL: NCT04987554
Title: Modulation of the Immune Response by AM3 Glycoconjugate.
Brief Title: Glycophosphopeptical AM3 A Potential Adjuvant in the Treatment of SARS-CoV-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valladolid (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Diego Fernandez Lazaro, Professor Doctor, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020.08.10
Record Dates: First submitted 2021-07-29; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19; AM3; treatment; immunomodulation
MeSH Terms: conditions — COVID-19 | interventions — Immunoferon

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AM3 supplementation group (Experimental): 2 capsules for 30 consecutive days, distributed in a single daily oral intake in the morning on an empty stomach.
  Interventions: Dietary Supplement: glycophosphopeptical AM3
- Control Group (Placebo Comparator): 2 capsules for 30 consecutive days, distributed in a single daily oral intake in the morning on an empty stomach.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: glycophosphopeptical AM3 — 3 g/day of AM3
  Other Names: Inmunoferon
  Arms: AM3 supplementation group
Other: Placebo — 3 g/day of placebo
  Arms: Control Group

SUMMARY:
Introduction: In late 2019, a novel human coronavirus was detected in Wuhan, China, causing an outbreak of the severe acute respiratory syndrome - Coronavirus 2 (SARS-CoV-2). The disease that SARS-CoV-2 causes was named coronavirus disease 2019 (COVID-19). The virus rapidly spread throughout China and beyond, causing a public health challenge of global concern. Today, the availability of safe and effective drugs to treat COVID-19 remains limited, and symptomatic supportive treatments are the foundations of care. A natural glycophosphopeptical, AM3 has been shown to effectively improve the progression of infectious respiratory diseases with no side effects. In this context, AM3 could maintain an adequate immune status and serve as a therapeutic tool against COVID-19.

Study Aim: The effect of AM3 supplementation on the progression of COVID-19 patients. To evaluate the existence of significant differences between control and intervention groups in the progression of severe COVID-19 disease.

Methods: Double-blind randomized controlled clinical trial in collaboration with the Health Care Management of Soria. At the start of the trial, eligible patients will be randomized in a 1:1 ratio into two intervention and control groups. Block randomization with participants based on gender will be used. 120 patients with a confirmed diagnosis of COVID-19 by PCR and/or antigen testing will be randomized to the control group (placebo treatment) or experimental group (AM3 treatment), respectively. Patients will be randomly divided into two groups, the AM3 supplementation group (n=60) and the control group (n=60). The intervention group will be administered 2 indistinct capsules of AM3 (3 g/day of AM3) for 30 consecutive days, distributed in a single daily oral intake in the morning on an empty stomach. The control group will be administered a placebo of identical appearance of 2 indistinct capsules for a single daily intake in the morning, same dose as the experimental group (3 g/day of placebo), for 30 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Males and females
* Confirmed clinical diagnosis of COVID-19 positive by Real-Time Reverse Transcription Polymerase Chain Reaction (RT-PCR) and/or SARS-CoV-2 Antigen Test performed 120 hours prior to patient inclusion in the study
* LDH 250-400 U/L
* Acceptance of informed consent signature
* IMC: 18.5-30
* Patients not participating in other trials
* No hepatic and renal disorders
* Possession of mental faculties to participate in the study

Exclusion Criteria:

* Patients with rare and specific viral diseases such as HIV
* Patients undergoing chemotherapy during the last 2 months
* Any other condition/pathology diagnosed by the medical specialist that prevents them from participating in the trial
* Intake of vitamin complexes or functional foods

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lactato deshidrogenasa (LDH) | 1day
  a catalytic enzyme found in many tissues of the body
Lactato deshidrogenasa (LDH) | 30 days
  a catalytic enzyme found in many tissues of the body

SECONDARY OUTCOMES:
Creatine kinase (CK) | 1day and 30 days
  CK is an enzyme expressed by various tissues and cell types.
Myoglobin (Mb) | 1day and 30 days
  Mb is a muscle heteroprotein
Aspartate Aminotransferase (AST) | 1day and 30 days
  markers of liver damage
Alanine Aminotransferase (ALT) | 1day and 30 days
  markers of liver damage
Interleukin 6 (IL-6) | 1day and 30 days
  inflammatory marker
Interleukin 1β (IL-1β) | 1day and 30 days
  inflammatory marker
tumor necrosis factor (TNF-α) | 1day and 30 days
  inflammatory marker
tumor necrosis factor receptor (TNFR-α) | 1day and 30 days
  inflammatory marker
C-reactive protein (CRP) | 1day and 30 days
  inflammatory marker; acute phase reactants.
Ferritin (FER) | 1day and 30 days
  Fer is a protein that stores iron in the cells; acute phase reactants - inflammatory marker

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud "La Milagrosa" Soria Sur, Soria, Spain

IPD SHARING:
Plan to Share IPD: Undecided